CLINICAL TRIAL: NCT05672329
Title: Functional Residual Capacity Under Apnoeic Oxygenation with Different Flow Rates in Children: a Single-centre Prospective Randomized Controlled Trial
Brief Title: Functional Residual Capacity Under Apnoeic Oxygenation with Different Flow Rates in Children
Acronym: FUTURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Riva (Other)
Responsible Party: Sponsor-Investigator, Thomas Riva, Prof. Dr. med., Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Fuchs-Riva2022
Record Dates: First submitted 2022-12-21; First posted 2023-01-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Apnea; Anesthesia; Intubation Complication; Children, Only; Apnea Infant; Atelectasis; Ventilation Therapy; Complications
Keywords: Atelectasis; Apnoeic oxygenation; High-flow nasal oxygen; Silent spaces; Functional residual capacity; Paediatric anaesthesia
MeSH Terms: conditions — Apnea; Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1: Low-flow apnoeic oxygenation (Experimental): Group 1) 0.2 L/kg/min using OptiFlow system by Fisher&Paykel and an oxygen inspiration concentration FiO2 of 1.0;
  Interventions: Other: 0.2 L/kg/min, FiO2 1.0 + continuous jaw thrust
- Group 2: High-flow apnoeic oxygenation (Experimental): Group 2) 2 L/kg/min using OptiFlow system by Fisher&Paykel and an oxygen inspiration concentration FiO2 of 1.0;
  Interventions: Other: 2 L/kg/min, FiO2 1.0 + continuous jaw thrust
- Group 3: Control group apnoeic oxygenation (Active Comparator): Group 3) 4 L/kg/min using OptiFlow system by Fisher&Paykel and an oxygen inspiration concentration FiO2 of 1.0;
  Interventions: Other: 4 L/kg/min, FiO2 1.0 + continuous jaw thrust
- Group 4: High-flow apnoeic oxygenation (Experimental): Group 4): 2 l/kg/min with OptiFlow FiO2 1.0 using OptiFlow-Switch system by Fisher&Paykel
  Interventions: Other: 2 L/kg/min using OptiFlow-Switch system, FiO2 1.0 + continuous jaw thrust

INTERVENTIONS:
Other: 0.2 L/kg/min, FiO2 1.0 + continuous jaw thrust — Apnoeic Oxygenation with flow rate 0.2 L/kg/min using OptiFlow system by Fisher&Paykel and an oxygen inspiration concentration FiO2 of 1.0
  Arms: Group 1: Low-flow apnoeic oxygenation
Other: 2 L/kg/min, FiO2 1.0 + continuous jaw thrust — Apnoeic Oxygenation with flow rate 2 L/kg/min using OptiFlow system by Fisher&Paykel and an oxygen inspiration concentration FiO2 of 1.0
  Arms: Group 2: High-flow apnoeic oxygenation
Other: 4 L/kg/min, FiO2 1.0 + continuous jaw thrust — Apnoeic Oxygenation with flow rate 4 L/kg/min using OptiFlow system by Fisher&Paykel and an oxygen inspiration concentration FiO2 of 1.0
  Arms: Group 3: Control group apnoeic oxygenation
Other: 2 L/kg/min using OptiFlow-Switch system, FiO2 1.0 + continuous jaw thrust — Apnoeic Oxygenation with flow rate 2 L/kg/min using OptiFlow-Switch system by Fisher&Paykel and an oxygen inspiration concentration FiO2 of 1.0
  Arms: Group 4: High-flow apnoeic oxygenation

SUMMARY:
During induction of general anaesthesia physiological breathing stops and needs to be artificially established with facemask ventilation, and finally tracheal intubation or placement of a supraglottic airway. During the airway management, when lungs are not or only poorly ventilated, there is a risk for atelectasis. These atelectasis can contribute to respiratory adverse events (e.g. pulmonary infection or respiratory insufficiency) during or after general anaesthesia. High-flow nasal oxygen (HFNO) is the administration of heated, humidified and blended air/oxygen mixture via a nasal cannula at rates ≥ 2 L/kg/min. HFNO used during airway management (i.e. intubation) can extend the tolerance for apnea, the time from end of physiological breathing until artificial ventilation is established. The main objective of this study is thus to investigate the variations of poorly ventilated lung units (i.e., silent spaces) as a surrogate for functional residual capacity measured by electrical impedance tomography to dynamically assess atelectasis formation and regression under apnoeic oxygenation with different flow rates.

DETAILED DESCRIPTION:
High-flow nasal oxygen (HFNO) is the administration of heated, humidified and blended air/oxygen via nasal cannula at rates ≥ 2 L/kg/min. HFNO is an open system that can be used with nasal prongs of different sizes and was developed in neonatal intensive care unit for preterm babies with apnoea as alternative to continuous positive airway pressure (CPAP). Due to its ease of use and safety to apply to a wide range of indication HFNO is increasingly gaining interest for providing respiratory support in paediatric patients and in adults in ICU with respiratory failure. In adult populations, the use of HFNO permits to prevent desaturation during tracheal intubation of intensive care patients with mild-to-moderate hypoxemia. An application for HFNO in adults and children, is the extension of safe apnoea in patients who were undergoing general anaesthesia for hypopharyngeal or laryngo-tracheal surgery. This method, the so-called safe apnoeic oxygenation, also prevents hypoxemia in children during intubation. By using this technique, Patel et al. demonstrated a significate prolongation of apnoea time and proposed a ventilatory effect, as these studies revealed a slower increase in pCO2 than physiologically was expected. In these studies, researchers compared their data to studies from the 1950-ies, where CO2 increase during apnoea was investigated. In contrast, the investigators' previous research projects with HFNO did not confirm the claimed ventilatory effect in children and adults.

Furthermore studies performed in spontaneously breathing neonates and adults have shown the ability of HFNO to generate some increase in pharyngeal pressure, which could explain the improvement of oxygenation despite prolongation of apnea time. The investigators' previous study on adult patients showed that a relevant increase of pressure was nearly absent while patient's mouth was open. Currently, there is no data on the physiological pressure that is generated in the subglottic airway in apneic children treated with HFNO. The traditional measurement of intratracheal pressure with a catheter in the trachea is considered to pose a risk in small children.

The main objective of this study is thus to investigate the variations of poorly ventilated lung units (i.e., silent spaces) as a surrogate for functional residual capacity measured by electrical impedance tomography to dynamically assess atelectasis formation and regression under apnoeic oxygenation with different flow rates.

Eligible children will receive premedication with Midazolam rectal/oral 0.5 mg/kg or Dexmedetomidine nasal 2 mcg/kg 30 minutes before the beginning of the procedure (local SOPs of the paediatric anaesthesia departments). Mandatory monitoring will consist of non-invasive peripheral oxygen saturation (SpO2), heartrate (HR), and non-invasive blood pressure (NIBP). An intravenous line for drugs injection will be placed.

After start of anaesthesia (="induction"), adequate face-mask ventilation will be established. The sealed envelope for randomisation will then be opened. Standard anaesthesia will be continued using of intravenous propofol. Anaesthetic depth will be assessed using NarcotrendTM (NarcotrendTM, Hannover, Germany), maintaining values between 40 and 60. Additional study related non-invasive monitoring: transcutaneous tcCO2 and O2 (ToscaTM, Radiometer, Neuilly-Plaisance, France) measurement, thoracic electrical impedance tomography (EIT, PulmoVista 500, Draeger, Luebeck, Germany) and NIRS (Niro-200NX (Hamamatsu, Tokyo, Japan). ECG, pulse-oximetry, blood pressure, Narcotrend (NarcotrendTM, Hannover, Germany), thoracic EIT will be measured continuously, starting before induction while spontaneous breathing and ending 1 minute after the recruitment-manoeuvre. All patients will receive neuromuscular blockade medication of 2 x ED95 (standard intubation dose) to facilitate airway management. Neuromuscular block will be assessed using train-of-four (TOF) monitoring (TOF-Watch, Organon Ltd, Dublin, Ireland). A TOF value of zero before apnoea start and throughout the whole procedure will be deemed essential.

After that one minute of pressure support mask ventilation (Pmax 20 cm H20) with a backup respiratory rate of 20/min, normalized at a volume of 6-8 ml.kg-1 with 100% oxygen and will be applied. The ventilation will be discontinued, and the child will be left apnoeic for 5 minutes receiving oxygen according to the randomisation.

Children will be randomized to receive three different flow rates of 100% oxygen, warmed and humidified with the OptiFlow device (Fisher&PaykelTM, Auckland, New Zealand):

* group 1): 0.2 l/kg/min + continuous jaw thrust
* group 2): 2 l/kg/min + continuous jaw thrust
* group 3): 4 l/kg/min + continuous jaw thrust (control group)
* Group 4): 2 l/kg/min with OptiFlow FiO2 1.0 using OptiFlow-Switch system by Fisher&Paykel.

The nostrils must not be occluded by the nasal cannula by more than 50%. The time until desaturation from SpO2 100% to SpO2 95% will be measured. A chest ultrasound at end of intervention after definitive airway management will prove that no pneumothorax developed during the procedure.

Break-up criteria during apnoea are: SpO2 below 95%, transcutaneous CO2 above 70 mmHg, or time of apnoea >5 minutes, a decrease of NIRS >30% from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent by legal guardian
* Paediatric patients undergoing elective surgery requiring general anaesthesia at the Bern University Hospital - Inselspital in Bern
* Child weight between 10-20kg
* American Society of Anesthesiology (ASA) physical status 1 & 2 (healthy child, no severe co-morbidities)

Exclusion Criteria:

* Known or suspected difficult intubation
* Oxygen dependency
* Congenital heart or lung disease
* Obesity BMI (kg/m2) >30
* High aspiration risk (requiring rapid sequence intubation).

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Total change in lung impedance | 5 Minutes
  The total change in lung impedance measured in silent spaces and end-expiratory lung impedance (EELI) by using electrical impedance tomography (EIT), normalized to the impedance amplitude during mechanical ventilation at 6-8 ml.kg-1 measured after 5 min of apnea compared to baseline measurement.
  Data given in percent (%) for silent spaces and delta EELI.

SECONDARY OUTCOMES:
Time until desaturation to SpO2 95% | 5 Minutes
  In case of desaturation within the predefined apnoea time: time (in seconds) until desaturation from peripheral saturation (SpO2) 100% to 95%, measured by peripheral pulse oximetry in percent (%).
Changes in transcutaneous CO2 | 5 Minutes
  Changes in transcutaneous carbon dioxide (tcCO2) in mmHg/min during apnoea time
Changes in brain oxygenation | 5 Minutes
  Changes in brain oxygenation measured by near infrared spectroscopy (NIRS) during apnoea time given in percent (%)
Changes in silent spaces and EELI after 1 min PSV | 5 Minutes
  The total change in lung impedance measured in silent spaces and end-expiratory lung impedance (EELI) by using electrical impedance tomography, normalized to the impedance amplitude during mechanical ventilation at 6-8 ml.kg-1 after induction and 1 minute of pressure supported ventilation with backup frequency (PSV) at 6-8 ml/kg.
  Data given in percent (%) for silent spaces and delta EELI.
Changes in silent spaces and EELI after airway management | 5 Minutes
  Changes in silent spaces and end-expiratory lung impedance (EELI) by using electrical impedance tomography after airway management (i.e. supraglottic airway or intubation).
  Data given in percent (%) for silent spaces and delta EELI.
Changes in silent spaces and EELI after recruitment manoeuvre | 5 Minutes
  Changes in silent spaces and end-expiratory lung impedance (EELI) by using electrical impedance tomography after recruitment manoeuvre and 1 minute of mechanical ventilation at 6-8 ml/kg.
  Data given in percent (%) for silent spaces and delta EELI.
Time to 25%, 50% and 75% of total change in lung impedance | 5 Minutes
  Time to 25%, 50% and 75% of total change in lung impedance by using electrical impedance tomography in seconds (s).

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Fuchs, M.D., Principal Investigator — Department of Anaesthesiology and Pain Medicine, Inselspital, Bern University Hospital,; Thomas Riva, M.D., Study Director — Department of Anaesthesiology and Pain Medicine, Inselspital, Bern University Hospital,
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Inselspital, Bern University Hospital, University of Bern, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lippuner R, Pellaud C, Huber M, Greif R, Disma N, Riva T, Fuchs A, Riedel T. Efficacy of a lung recruitment manoeuvre in children undergoing general anaesthesia with a supraglottic airway. Br J Anaesth. 2025 Nov;135(5):1537-1542. doi: 10.1016/j.bja.2025.08.016. Epub 2025 Sep 23. PMID 40993003